CLINICAL TRIAL: NCT06954870
Title: Is Ozone Therapy an Effective Treatment for Lipedema? Comparison of Systemic and Local Ozone Treatments
Brief Title: Effect of Systemic and Local Ozone Therapy in Lipedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Başak Mansız-Kaplan, Assoc. Prof. Dr. Başak Mansız Kaplan Ankara Etlik City Hospital, Department of Physical Medicine and Rehabilitation, Head of the Orthopedic Rehabilitation Clinic, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/16
Record Dates: First submitted 2025-03-26; First posted 2025-05-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Lipedema; Pain; Activities of Daily Living; Musculoskeletal Ultrasound
MeSH Terms: conditions — Lipedema; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Systemic ozone therapy (Experimental): 1 session of 40 gamma per week, a total of three weeks of major ozone therapy will be applied
  Interventions: Other: Ozone therapy
- Local ozone therapy (Experimental): 10 gamma local ozone injection per week, a total of three weeks will be performed 5 times with 1 cm intervals to the painful points of the patient.
  Interventions: Other: Ozone therapy
- Both systemic and local ozone therapy (Experimental): 1 session of 40 gamma per week, a total of three weeks of major ozone therapy will be applied and also 10 gamma local ozone injection per week, a total of three weeks will be performed 5 times with 1 cm intervals to the painful points of the patient.
  Interventions: Other: Ozone therapy

INTERVENTIONS:
Other: Ozone therapy — As detailed in the research arms, major ozone application and local ozone application will be performed.

SUMMARY:
Lipedema is a disease characterized by enlargement of the subcutaneous tissue and is observed only in the female population. Recently, the inflammatory cascade has been suggested to be the initiator of lipoedema and to play a role in its progression. The presence of pain in the involved areas is the most important symptom affecting the patient's QoL.

In the literature, ozone therapy is used both locally and systemically in many diseases in which inflammation is involved in the etiopathogenesis. There are many studies on plantar fasciitis, lateral epicondylitis, rheumatoid arthritis, osteoarthritis, etc. In addition to its anti-inflammatory properties, ozone therapy, which has analgesic and aseptic properties, has not been found in the literature in patients with lipedema.

The aim of this study was to investigate the effect of ozone therapy on pain symptoms and subcutaneous tissue thickness in patients with lipedema and to compare local and systemic ozone applications in these patients.

DETAILED DESCRIPTION:
The study, which is planned as a prospective randomized intervention, will include 50 female patients aged 18-65 years with a diagnosis of lipedema by a physician who applied to Etlik City Hospital Physical Medicine and Rehabilitation clinic and had pain >4 evaluated by VAS.

Since there is no study evaluating ozone therapy in lipedema in the literature, the sample size calculated with G*Power 3.0.10a based on another ozone therapy study was found to be 15 patients each. Considering the possibility of dropout from the study, the sample size was determined as 50 volunteers in total.

After clinical diagnosis, pain with visual analog scale (VAS) and pain detect pain questionnaire will be applied to evaluate neuropathic pain. In patients with lipedema, measurements will be made by a physical medicine and rehabilitation physician with 10 years of experience in musculoskeletal ultrasonography from the areas previously defined ultrasonographically in the literature (Midpoint between the superior anterior iliac crest and the inferior patellar border, medial tubercle of the femur, midpoint between the tibial tuberosity and the medial malleolus, midpoint between the lateral malleolus and the fibular head, medial supramalleolar) with the ultrasonography device available in the clinic.Patients' age, comorbidities, medications and routine laboratory parameters such as neutrophil/lymphocyte ratio, platelet distribution width, mean platelet volume, sedimentation, CRP, hemogram values will be recorded. VAS, pain detection and ultrasonographic measurements will be repeated at the 1st and 3rd month after the end of the application.

After the patients were randomized into three groups, the first group will receive local ozone, the second group will receive systemic ozone, and the third group will receive both local and systemic ozone. Local ozone will be injected into the painful points of the patient at the level of the medial tubercle of the femur, 10 gamma 10 cc ozone injection will be made radiationally from 5 regions with 1 cm intervals under the guidance of USG (3 sessions). Systemic ozone application will be given in 3 sessions of 40 gamma each.

ELIGIBILITY:
Inclusion Criteria:

* To have been diagnosed with clinical lipedema.
* Pain assessed by VAS of 5 or more
* Being a woman
* Being between 18-65 years old

Exclusion Criteria:

* Presence of venous insufficiency leading to subcutaneous changes
* Having diseases that may cause edema
* Use of painkillers (NSAIDs/Opioids) up to 1 week before the injection
* Open wound or infection at the site of infection
* Bleeding disorders or use of anticoagulant, antiplatelet drugs uncontrolled systemic disease
* G6PD deficiency
* Cases where the pain cannot be explained by lipoedematous tissue

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lipedema is a disease that almost always affects women.
Enrollment: 45 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | before application, at 1st and 3rd month
  A visual analog scale will be used to assess pain intensity. In this scale, which is scored between 1-10, 0 indicates the best condition and 10 indicates the most severe pain.

SECONDARY OUTCOMES:
painDETECT Questionnaire | before application, at 1st and 3rd month
  painDETECT Questionnaire will be performed for neuropathic pain. A total score of 19 or more is indicative of likely neuropathic pain.
Subcutaneous ultrasonographic measurement | before application, at 1st and 3rd month
  Subcutaneous ultrasonographic measurement will be performed. The measurement of subcutaneous adipose tissue will be recorded in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Mansız Kaplan, MD,AssocProf, Principal Investigator — Ankara Etlik City Hospital, Department of Physical Medicine and Rehabilitation
Locations (1):
- Ankara Etlik City Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No